CLINICAL TRIAL: NCT06653244
Title: Morphine, Midazolam and Dexmedetomidine in the Management of Acute Cardiogenic Pulmonary Edema, Safety and Efficacy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Amany Said Abdel Haleem, Lecturer of Anesthesia and Intensive care, Menoufia University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 32024ANET10
Record Dates: First submitted 2024-10-13; First posted 2024-10-22 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2024-10

CONDITIONS: Sedative Adverse Reaction
MeSH Terms: interventions — Injections; Morphine; Midazolam

STUDY DESIGN:
Intervention Model Description: The patients will be randomized in a 1:1:1 ratio, (group Mi) midazolam (administered intravenously at a dosage of 1 mg, up to a maximum dose of 3 mg) [14], [15],(group Mo) morphine (administered intravenously at a dosage of 2-4 mg, up to a maximum dose of 8 mg [14], [15],(group Dex.) dexmedetomidine ( administered intravenously, Load: 0.25 mcg/kg IV over 10 minutes , Maintenance 0.2-0.7 mcg/kg/hr continuous IV 7 infusion according to haemodynamics and sedation score of patient ; not to exceed 24 hr
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- group Midazolam (Active Comparator): midazolam (administered intravenously at a dosage of 1 mg, up to a maximum dose of 3 mg) on demand
  Interventions: Drug: Injection
- GROUP Morphine (Active Comparator): morphine (administered intravenously at a dosage of 2-4 mg, up to a maximum dose of 8 mg every 12 hours
  Interventions: Drug: Injection
- Group Dexmedetomidine (Active Comparator): dexmedetomidine ( administered intravenously, Load: 0.25 mcg/kg IV over 10 minutes , Maintenance 0.2-0.7 mcg/kg/hr continuous IV 7 infusion according to haemodynamics and sedation score of patient ; not to exceed 24 hr
  Interventions: Drug: Injection

INTERVENTIONS:
Drug: Injection — dexmedimidine infusion
  Other Names: morphine injection; midazolam injection

SUMMARY:
Acute cardiogenic pulmonary edema is a stressful scenario with progressive respiratory failure that may lead to cardiorespiratory collapse within hours, or minutes unless therapeutic action is taken As the initial events in involve hemodynamic pulmonary congestion with high capillary pressures, diuretics, non-invasive ventilation (NIV) and vasodilators constitute the key armamentarium for the initial treatment.

DETAILED DESCRIPTION:
The patients will be randomized in a 1:1:1 ratio, (group midazolam i) midazolam (administered intravenously at a dosage of 1 mg, up to a maximum dose of 3 mg) (group morphine) morphine (administered intravenously at a dosage of 2-4 mg, up to a maximum dose of 8 mg [14], [15],(group Dexmedetomidine.) dexmedetomidine ( administered intravenously, Load: 0.25 mcg/kg IV over 10 minutes , Maintenance 0.2-0.7 mcg/kg/hr continuous IV infusion according to haemodynamics and sedation score of patient ; not to exceed 24 hr

• Boluses of morphine, midazolam and dexmeddetomidine will be repeated on demand according to Ramsay sedation scale.

• All patients will be assessed for need of noninvasive ventilation by total face mask connected to ventilator.

• Medical therapy with intravenous boluses of loop diuretics, intravenous infusions of nitroglycerine, oxygen supplementation will be provided by physicians according to their clinical judgment

• The target in all patients is to provide anxiolytic or light sedation effect for good compliance to noninvasive ventilation and reducing of pulmonary congestion.

• The expected sedation scores (Ramsay score 2-3) will be achieved in all of the patients taking morphine, midazolam or dexmedetomidine

ELIGIBILITY:
Inclusion Criteria:

* Age >18 year with a clinical diagnosis of ACPE with severe dyspnea and anxiety.
* Patients able to verbally acknowledge the risks in receiving midazolam, morphine or dexmedetomidine.-

Diagnosis of ACPE was defined by the association of sudden onset of dyspnoea, the presence of bilateral rales on auscultation, respiratory rate >25 breaths/min and pulse oxygen saturation <90% in room air. diagnosis will be confirmed by echocardiography and lung ultrasound

Exclusion Criteria:

* Patients with history of asthma, severe stenotic valvular disease. • Cardiovascular collapse or an impaired level of consciousness (Glasgow Coma Scale score of ≤8 points).

Immediate indication for intubation.

• Suspicion of ST-segment elevation, acute coronary syndrome needing interventions.

• Known severe liver or renal disease, pneumonia, poor chance of survival due to a pre-existing condition.

• Psychiatric disorders.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Clinical improvement in length of hospital stay | 48 hours

SECONDARY OUTCOMES:
In- hospital all- cause mortality. | 72 hours
mortality | 30-day

CONTACTS AND LOCATIONS:
Locations (1):
- Menofia university, Shibīn al Kawm, Menofia, Egypt